CLINICAL TRIAL: NCT04693702
Title: Observational Study of Vision Improvement in Patients With Retinal Disorders
Status: Completed | Type: Observational
Sponsor: Optimal Acuity Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Retro2
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Age-related Macular Degeneration; Diabetic Macular Edema
Keywords: Age-related macular degeneration; Diabetic macular edema
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Age-related Macular Degeneration
  Interventions: Device: Corneal treatment by a low vision aid device
- Diabetic Macular Edema
  Interventions: Device: Corneal treatment by a low vision aid device

INTERVENTIONS:
Device: Corneal treatment by a low vision aid device — Near infrared light is used to irradiate the cornea to change the modulus of small volumes of anterior stroma. The modulus change produces a change in light distribution onto the retina. Light rays are redirected from dysfunctional areas of the retina to functional areas, thereby improving patient vision.

SUMMARY:
The purpose of this study is to assess the vision improvement achieved by patients with retinal disorders who received corneal treatments by a low vision aid device.

DETAILED DESCRIPTION:
The purpose of this study is to assess the vision improvement achieved by patients with retinal disorders, including age-related macular degeneration and diabetic macular edema, who received corneal treatments by a low vision aid device. Patient records will be analyzed to determine measures of vision improvement including best spectacle-corrected distance visual acuity (CDVA). Analyses will include descriptive statistics and correlation between outcomes and baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. - Female or male
2. - Any race
3. - Patient is at least 50 years old
4. - Patient has diagnosed retinal disorder that causes central vision loss in one or both eyes
5. - Treated eyes, at time of treatment, were pseudophakic or phakic with no significant vision loss due to cataract
6. - Patient had moderate to severe baseline vision impairment with CDVA of 20/63 or worse (decimal = 0.317 or less; logMAR greater than or equal to 0.50) in the treated eye(s)
7. - Patient CDVA records are available at baseline and at 1m or longer post-Tx times

Exclusion Criteria:

1 - Corneal disease or disorder in either eye 2 - Increased intraocular pressure (above 20mm Hg), glaucoma or history of glaucoma 3 - Presence or history of any other condition or finding that, in the opinion of the investigator, makes the patient unsuitable for retrospective observational study

-

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with vision impairment due to retinal disorders involving central vision loss
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
CDVA | 12 months
  Best spectacle-corrected distance visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Berry, PhD, Principal Investigator — Optimal Acuity Corporation
Locations (1):
- Bochner Eye Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No